CLINICAL TRIAL: NCT03168178
Title: A Randomized Trial in Intrapartum Fever Of No Antibiotics for Low-risk Women (RATIONAL)
Brief Title: Intrapartum Fever: Antibiotics Versus no Treatment
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Participant enrollment was much more challenging than anticipated.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Heather Campbell, Principal Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 91955
Record Dates: First submitted 2017-05-18; First posted 2017-05-30 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Chorioamnionitis; Intrapartum Fever; Intra-amniotic Infection
MeSH Terms: conditions — Chorioamnionitis

STUDY DESIGN:
Intervention Model Description: Low risk women will be randomized to standard antibiotic treatment versus no antiobiotics.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Antibiotic Treatment (Active Comparator): Standard antibiotic treatment provided to patient. Placenta submitted for pathologic exam. Maternal and neonatal outcomes collected.
  Interventions: Drug: Standard Antibiotic Treatment
- No Antibiotic Treatment (Experimental): No Antibiotic treatment given. Placenta submitted for pathologic exam. Maternal and neonatal outcomes collected.
  Interventions: Other: No Antibiotic Treatment

INTERVENTIONS:
Drug: Standard Antibiotic Treatment — Participants randomized to this intervention will receive standard antibiotic treatment.
  The placenta will be submitted for pathologic exam after delivery and investigators will collect maternal and neonatal outcomes
  Arms: Standard Antibiotic Treatment
Other: No Antibiotic Treatment — Participant randomized to this arm of the study will not receive antibiotics. The placenta will be submitted for pathologic exam after delivery and investigators will collect maternal and neonatal outcomes
  Arms: No Antibiotic Treatment

SUMMARY:
The purpose of this study is to determine whether antibiotics can be safely avoided in women who develop a fever during labor. Because investigators have no accurate tests to determine whether women who develop fever during labor have intra-amniotic infection, antibiotics are often used to prevent spread of infection to the fetus.

DETAILED DESCRIPTION:
A fever > 100.4 F during labor (intrapartum fever) complicates up to 14% of term deliveries, and is commonly considered a sign of intrauterine infection. Despite studies showing that most causes of maternal intrapartum fever are non-infectious, intrapartum fever often prompts the diagnosis of chorioamnionitis/intrauterine infection, or what is now known as 'triple I' (intra-amniotic infection or inflammation). Diagnosis of triple I is primarily based on clinical findings such as maternal fever, maternal leukocytosis, uterine tenderness, foul-smelling or purulent amniotic fluid, and fetal tachycardia. A minimum of two of these criteria for diagnosis, although this distinction is somewhat artificial as fetal tachycardia is highly associated with maternal fever. The poor performance of clinical signs and lack of effective biomarkers to identify neonatal infection results in over treatment of both mothers and infants.

Avoiding antibiotic use in mothers and infants is desirable in order to avoid unnecessary separation after birth, decreasing cost and interventions in newborns, and to avoid altering the infant's microbiome (the bacteria newborns carry on their skin, mucosal membranes, and in their gut at the time of birth). Infants with altered microbiomes may be at risk for skin, pulmonary, and gastrointestinal disorders. The investigators in this trial are randomizing women with fever during labor who are felt to be a low risk for true infection to antibiotic treatment compared to no antibiotics in order to determine if antibiotics can be safely avoided for these women and their infants.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 34-42 weeks gestation
* Singleton fetus
* Admitted for labor management & develops a fever of 100.4 F or greater

Exclusion Criteria:

* Known fetal anomaly
* Other indication for intrapartum antibiotics (endocarditis prophylaxis, other known maternal infection)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
Neonatal antibiotic treatment as recommended by the EONS (Early Onset Neonatal Sepsis) calculator. | Within 2 hours of delivery
  All newborns will have a screening assessment including physical exam and vital signs, and this data along with maternal and delivery data is entered into the Kaiser Permanente Early Onset Neonatal Sepsis (EONS) calculator. The EONS calculator estimates the risk of sepsis and recommends observation, additional evaluation, or empiric antibiotic treatment.

SECONDARY OUTCOMES:
Positive blood culture | Up to 4 days after birth
  For infants who have a blood culture obtained by recommendation of the EONS calculator, the presence of significant bacterial growth will be considered a positive culture.
Need for NICU admission | Up to 4 weeks after birth
  Admission of the infant to the Newborn Intensive Care Unit
Newborn length of stay | Up to 4 weeks after birth
  Days hospitalized after birth
Maternal endometritis | Up to 4 weeks after birth
  The diagnosis of endometritis made by the patient's OB provider requiring treatment with antibiotics.
Maternal length of stay | Up to 4 weeks after birth
  Days hospitalized after delivery
Patient satisfaction | 6-8 weeks after delivery
  Satisfaction with maternal and newborn care using a standardized survey administered by phone at 6-8 weeks after delivery
Cost | Up to 4 weeks after birth
  The hospital charges for mother and infant

CONTACTS AND LOCATIONS:
Overall Officials: Heather Campbell, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Department of Obstetrics & Gynecology, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smulian JC, Bhandari V, Vintzileos AM, Shen-Schwarz S, Quashie C, Lai-Lin YL, Ananth CV. Intrapartum fever at term: serum and histologic markers of inflammation. Am J Obstet Gynecol. 2003 Jan;188(1):269-74. doi: 10.1067/mob.2003.11. PMID 12548228
- [Background] Smulian JC, Shen-Schwarz S, Vintzileos AM, Lake MF, Ananth CV. Clinical chorioamnionitis and histologic placental inflammation. Obstet Gynecol. 1999 Dec;94(6):1000-5. doi: 10.1016/s0029-7844(99)00416-0. PMID 10576190
- [Background] Roberts DJ, Celi AC, Riley LE, Onderdonk AB, Boyd TK, Johnson LC, Lieberman E. Acute histologic chorioamnionitis at term: nearly always noninfectious. PLoS One. 2012;7(3):e31819. doi: 10.1371/journal.pone.0031819. Epub 2012 Mar 7. PMID 22412842
- [Background] Taylor JA, Opel DJ. Choriophobia: a 1-act play. Pediatrics. 2012 Aug;130(2):342-6. doi: 10.1542/peds.2012-0106. Epub 2012 Jul 9. PMID 22778303
- [Background] Escobar GJ, Puopolo KM, Wi S, Turk BJ, Kuzniewicz MW, Walsh EM, Newman TB, Zupancic J, Lieberman E, Draper D. Stratification of risk of early-onset sepsis in newborns >/= 34 weeks' gestation. Pediatrics. 2014 Jan;133(1):30-6. doi: 10.1542/peds.2013-1689. Epub 2013 Dec 23. PMID 24366992
- [Background] Cuna A, Hakima L, Tseng YA, Fornier B, Islam S, Quintos-Alagheband ML, Khullar P, Weinberger B, Hanna N. Clinical dilemma of positive histologic chorioamnionitis in term newborn. Front Pediatr. 2014 Apr 4;2:27. doi: 10.3389/fped.2014.00027. eCollection 2014. PMID 24772410
- [Background] Evers AC, Nijhuis L, Koster MP, Bont LJ, Visser GH. Intrapartum fever at term: diagnostic markers to individualize the risk of fetal infection: a review. Obstet Gynecol Surv. 2012 Mar;67(3):187-200. doi: 10.1097/OGX.0b013e31824bb5f1. PMID 22901952
- [Background] Buhimschi IA, Christner R, Buhimschi CS. Proteomic biomarker analysis of amniotic fluid for identification of intra-amniotic inflammation. BJOG. 2005 Feb;112(2):173-81. doi: 10.1111/j.1471-0528.2004.00340.x. PMID 15663581
- [Background] Stoll BJ, Hansen NI, Sanchez PJ, Faix RG, Poindexter BB, Van Meurs KP, Bizzarro MJ, Goldberg RN, Frantz ID 3rd, Hale EC, Shankaran S, Kennedy K, Carlo WA, Watterberg KL, Bell EF, Walsh MC, Schibler K, Laptook AR, Shane AL, Schrag SJ, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Early onset neonatal sepsis: the burden of group B Streptococcal and E. coli disease continues. Pediatrics. 2011 May;127(5):817-26. doi: 10.1542/peds.2010-2217. Epub 2011 Apr 25. PMID 21518717
- [Background] Newman TB, Puopolo KM, Wi S, Draper D, Escobar GJ. Interpreting complete blood counts soon after birth in newborns at risk for sepsis. Pediatrics. 2010 Nov;126(5):903-9. doi: 10.1542/peds.2010-0935. Epub 2010 Oct 25. PMID 20974782